CLINICAL TRIAL: NCT01889368
Title: Effect of a Grape Seed Extract (GSE) on Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Illinois Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 329493; 329493-4 (Other: UC Davis)
Record Dates: First submitted 2012-10-10; First posted 2013-06-28 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Metabolic Syndrome
Keywords: Insulin resistance; Central adiposity; Elevated blood pressure; Vascular reactivity; Elevated triglycerides; Low high-density lipoprotein (HDL)
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Obesity, Abdominal; Hypertension; Hypertriglyceridemia | interventions — Grape Seed Extract; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grape Seed Extract (Active Comparator): This is a 30 day arm. At the baseline study visit, subjects will consume one 300 mg capsule of MegaNatural Gold followed by 3 high fat meals: breakfast, lunch, and dinner. Blood will be drawn at specified intervals throughout the day. Flow mediated dialysis will be performed before breakfast and again 1.5 hours later, after capsule consumption and breakfast. A minimum 14 day washout period will be between arms if this is the first arm in the randomized cross-over.
  Interventions: Dietary Supplement: Grape Seed Extract
- Placebo (Placebo Comparator): This is a 30 day arm. At the baseline study visit, subjects will consume one placebo (maltodextrin) capsule followed by 3 high fat meals: breakfast, lunch, and dinner. Blood will be drawn at specified intervals throughout the day. Flow mediated dialysis will be performed before breakfast and again 1.5 hours later, after capsule consumption and breakfast. A minimum 14 day washout period will be between arms if this is the first arm in the randomized cross-over.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Grape Seed Extract — 300 mg capsule of Grape Seed Extract; 1 capsule will be consumed for an acute post-prandial study day and 1 capsule will be consumed daily for 30 days.
  Other Names: MegaNatural Gold
  Arms: Grape Seed Extract
Dietary Supplement: Placebo — 300 mg capsule of maltodextrin; 1 capsule will be consumed for an acute post-prandial study day and 1 capsule will be consumed daily for 30 days.
  Other Names: Maltodextrin
  Arms: Placebo

SUMMARY:
In people with the metabolic syndrome, the investigators hypothesize that administration of a single 300 mg dose of a grape seed extract (GSE) will reduce insulin resistance (how well cells in the body can take up and use glucose), oxidative stress, and the amount of oxidized LDL in the blood during a 24 hour period. These measurements will be assessed at hourly intervals during the 24 hour study day protocol. Additionally, the investigators hypothesize that daily administration of 300 mg of GSE for 30 days will decrease baseline insulin resistance, oxidative stress, and the level of oxidized LDL in the blood.

DETAILED DESCRIPTION:
In people with the metabolic syndrome, the investigators hypothesize that administration of a single 300 mg dose of a grape seed extract (GSE) will reduce insulin resistance (how well cells in the body can take up and use glucose), oxidative stress, and the amount of oxidized LDL in the blood during a 24 hour period. Each of these can be elevated after eating high fat meals, which are commonly found in the average Western diet. To better assess the impact of these high fat eating patterns, three standardized high fat meals will be served during the study day: breakfast, lunch, and dinner. Measurements in the blood will be assessed at hourly intervals during the 24 hour study day protocol. Additionally, the investigators hypothesize that daily administration of 300 mg of GSE for 30 days will decrease baseline insulin resistance, oxidative stress, and the level of oxidized LDL in the blood when this 24 hour study day protocol is repeated and breakfast, lunch, and dinner are again served.

Insulin resistance will be measured using a comparison of insulin and glucose levels in the blood. Oxidative stress, a measure of inflammation, will be measured by cytokines levels in the blood. The level of oxidized LDL will be measured in the blood. The investigators also plan to undertake a subsidiary pharmacokinetic study on the various polymers which are known to be present in grape seed extracts to determine their bio-availability and their relationship to the biological effects observed.

ELIGIBILITY:
Inclusion Criteria

* Metabolic Syndrome, based on subject meeting at least 3 of the following criteria:
* Abdominal obesity with waist circumference > 40 inches in men or > 35 inches in women,
* Pre-hypertension with blood pressure > 135/85,
* Fasting blood glucose levels above 110 mg/dl,
* Plasma triglyceride levels in excess of 150 mg/dl,
* HDL levels below 40 mg/dl in men or 50 mg/dl in women.

Exclusion Criteria:

* Any known systemic disease,
* Diabetes,
* Alcohol consumption > 1-2 drinks/week,
* Taking any medications or supplements that will affect metabolism, their ability to exercise or oxidative status,
* Smokers,
* Female subjects having abnormal menstrual cycles, taking oral contraceptives, pregnant or lactating.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Changes in insulin resistance | Baseline and 30 days
  Insulin resistance will be assessed by comparing the baseline fasting insulin concentration to the fasting insulin concentration after intervention period of 30 days; the Homeostatic Model Assessment (HOMA) value will be utilized for comparisons.

SECONDARY OUTCOMES:
Changes in oxidized LDL (oxLDL) concentrations | Baseline and 24 hour post-prandial response
  Changes in oxLDL concentrations will be assessed by ELISA methodology. Changes in the 24 hour post-prandial response will be assessed at one hour intervals during the post-prandial study days, after capsule consumption and eating 3 high fat meals.
Changes in oxidative stress | Baseline and 24 hour post-prandial response
  Changes in the 24 hour post-prandial oxidative stress response will be assessed at one hour intervals during the post-prandial study days, after capsule consumption and eating 3 high fat meals. Changes in oxidative stress will be assessed by measuring cytokine production using ELISA methodology.
Changes in vascular stress | Baseline and 1 hour post-prandial
  Changes in oxidative stress will be assessed by flow mediated dialysis (FMD). Changes will be assessed at baseline and one hour after capsule consumption and eating a high fat breakfast meal.
Changes in insulin response | Baseline and 24 hour post-prandial response
  Changes in the 24 hour post-prandial insulin response will be assessed at one hour intervals during the post-prandial study days, after capsule consumption and eating 3 high fat meals.
Changes in oxidized LDL (oxLDL) concentrations | Baseline and 30 days
  Changes in oxLDL concentrations will be assessed by ELISA methodology. Changes in the 24 hour post-prandial response will be assessed at one hour intervals during the post-prandial study days, after capsule consumption and eating 3 high fat meals. The response from the baseline visit will be compared to the response obtained during the day 30 visit.
Changes in insulin response | Baseline and 30 days
  Changes in the 24 hour post-prandial insulin response will be assessed at one hour intervals during the post-prandial study days, after capsule consumption and eating 3 high fat meals. The response from the baseline visit will be compared to the response obtained during the day 30 visit.
Changes in oxidative stress | Baseline and 30 days
  Changes in the 24 hour post-prandial oxidative stress response will be assessed at one hour intervals during the post-prandial study days, after capsule consumption and eating 3 high fat meals. Changes in oxidative stress will be assessed by measuring cytokine production using ELISA methodology. The response from the baseline visit will be compared to the response obtained during the 30 day visit.
Changes in vascular stress | Baseline and 30 days
  Changes in oxidative stress will be assessed by flow mediated dialysis (FMD). Changes will be assessed at baseline and one hour after capsule consumption and eating a high fat breakfast meal. Results obtained during the first post-prandial study visit will be compared to those obtained 30 days later.

CONTACTS AND LOCATIONS:
Overall Officials: Chulani T Kappagoda, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- VA Hospital, Mather, Mather, California, United States